CLINICAL TRIAL: NCT01611506
Title: Integration of Cetuximab, in Combination With Local Radiotherapy, in Perioperative Chemotherapy of Resectable and Locally Advanced Gastric Cancer. A Pilot Phase Ib-trial
Brief Title: Combination Chemotherapy, Cetuximab and Radiation for Patients With Localized Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Outcome of EXPAND study (no benefit from adding cetuximab to the first-line chemotherapy in advanced gastric cancer in the overall patient population)
Sponsor: Dr Anna Dorothea Wagner (Other)
Responsible Party: Sponsor-Investigator, Dr Anna Dorothea Wagner, Médecin associée, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-CePO-B354re (gastric)
Record Dates: First submitted 2012-05-15; First posted 2012-06-05 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab, capecitabine, cisplatin based chemoradiation (Experimental): Induction chemotherapy:
  3 cycles (of 3 weeks) with capecitabine, cisplatin and weekly cetuximab: Cetuximab 400mg/m2 (loading dose)on day 1 and 250mg/m2 weekly thereafter, Cisplatin 80mg/m2 on day 1 every three weeks, Capecitabine 1000mg/m2 twice daily from the evening of day 1 to the morning of day 15 within each 3 weeks cycle.
  Followed by:
  Radio-chemo-immunotherapy:
  Cetuximab 250mg/m2 weekly on day 1, Cisplatin 30mg/m2 weekly on day 1, Radiotherapy (dose escalation levels) 36/39.6/45 Gy(according to dose level) in 5 fractions of 1.8 Gy per week
  Surgery:
  Will be performed 4-6 weeks after neoadjuvant radiochemotherapy
  Postoperative treatment:
  3 cycles of Chemo-immunotherapy with cetuximab, cisplatin and capecitabine -as described above- will be administered postoperatively if the patient has recovered adequately from surgery and the treatment is considered as feasible by the investigator.
  Interventions: Biological: Cetuximab; Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Cetuximab — Induction chemotherapy:
  Cetuximab 400mg/m2 (loading dose) on day 1 Cetuximab 250mg/m2 weekly thereafter
  Followed by:
  Cetuximab 250mg/m2 weekly on day 1 during chemoradiation
  Postoperative treatment:
  3 cycles of Cetuximab 250mg/m2 weekly on day 1
Drug: Capecitabine — Induction chemotherapy:
  Capecitabine 1000mg/m2 twice daily from the evening of day 1 to the morning of day 15 within each 3 weeks cycle
  Postoperative treatment:
  Capecitabine 1000mg/m2 twice daily from the evening of day 1 to the morning of day 15 within each 3 weeks cycle
Drug: Cisplatin — Induction chemotherapy:
  Cisplatin 80mg/m2 on day 1 of each 21 day cycle
  Followed by:
  Cisplatin 30mg/m2 weekly on day 1 during chemoradiation
  Postoperative treatment:
  Cisplatin 80mg/m2 on day 1 of each 21 day cycle

SUMMARY:
RATIONALE: Radiotherapy is currently the most efficient way to induce pathologic responses, which are associated with a favorable prognosis in localized tumors. Novel radiotherapy techniques are associated with significantly less toxicity than traditional radiation protocols and permit to avoid the toxicity to adjacent organs. Established chemotherapy regimens, such as cisplatin and capecitabine, and monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Giving radiation therapy together with cisplatin and cetuximab before surgery aims to induce a pathological response and improve the prognosis after surgery.

PURPOSE: This phase I trial is studying the side effects and best dose of radiation therapy when given together with cisplatin and cetuximab in treating patients who are undergoing surgery for locally advanced gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

• To determine the maximum tolerated dose of radio-chemo-immunotherapy - in patients with localized or locally advanced gastric cancer

Secondary

* To determine the efficacy, as measured by major histopathological response rates (tumor regression grade 1 and 2)
* Metabolic response
* Secondary resectability
* R-0 resection rate
* Surgical morbidity
* Toxicity
* Overall survival
* Time to local and systemic progression after R0-resection
* Feasibility

OUTLINE: Prospective, multicenter, open-label dose escalating phase Ib trial

During induction chemo-immuno-therapy, patients receive cetuximab IV over 1-2 hours on days 1, cisplatin IV over 1 hour on day 1 and capecitabine twice daily per os from the evening of day 1 to the morning of day 15. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Radiotherapy will start after the end of the third cycle of chemotherapy and be performed concomitantly with weekly cetuximab and cisplatin.

Cohorts of 3-6 patients receive escalating doses of radiotherapy (levels of 36/39.6/45 Gy) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which maximum 3 of 12 patients experience dose-limiting toxicity.

Gastric resection should be performed within 4-6 weeks after completion of neoadjuvant treatment.

4-6 weeks after surgery, a further 3 cycles of chemo-immuno-therapy will be administered if the patient has recovered from surgery and the treatment is considered as feasible by the investigator.

For note: Cisplatin may be replaced by oxaliplatin during induction chemotherapy and postoperative chemotherapy. In case if oxaliplatin is used to replace cisplatin during induction chemotherapy, replacement of cisplatin by oxaliplatin during radio-chemo-immunotherapy may also be considered by the investigator.

Capecitabine may be replaced by infusional 5-FU on day 1-5 every 21 days in case of contraindications to capecitabine.

In case if both cisplatin and capecitabine are to be replaced, 4 cycles of FOLFOX-6 (d-l leucovorin, followed by 5-FU bolus and a continuous infusion of over 46 hours every 2 weeks should be administered in combination with cetuximab).

Patients undergo tumor tissue and blood sample collection periodically for biological studies. Samples are analyzed for major histopathological response.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, localized (UICC stage I-II, T1-2, N1-2 or T3N0) or locally advanced (UICC stage III, T3-4, N+) gastric or Siewert Type II and III GE-junction adenocarcinoma. Tumor stage is determined by thoraco-abdominal CT-scan, EUS, as well as mandatory laparoscopy to rule out peritoneal carcinomatosis within 28 days prior to registration.
* ECOG-status 0-1
* Hematologic, liver, and renal function normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment

Exclusion Criteria:

* Peritoneal carcinomatosis, as diagnosed by mandatory laparoscopy or distant metastasis
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, or treatment within a clinical trial within 30 days prior to trial entry
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, no myocardial infarction within the last 12 months, unstable angina pectoris, or significant arrhythmia)
* Active or uncontrolled infection.
* Definitive contraindications for the use of corticosteroids as premedication
* Prior systemic (chemo- or targeted) treatment. Prior radiotherapy to the upper abdomen
* Any contraindication to treatment with cetuximab, capecitabine or cisplatin
* Any concomitant medication which is contraindicated for use with the trial drugs, such as sorivudin or brivudin
* HER-2 over expression, as determined by immunohistochemistry (IHC 3+) or the combination of IHC and FISH (IHC 2+/FISH+)
* Previous malignancy within 5 years, with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Known hypersensitivity against any of the study drugs (cetuximab, cisplatin or capecitabine) or any component of the trial drugs
* Known deficit of dihydropyrimidine dehydrogenase
* Pre-existing peripheral neuropathy > grade I
* Due to known interactions of coumarin antagonists (e.g. warfarin) and capecitabine patients requiring oral anticoagulation should be included in the study only after a switch from oral anticoagulation to low molecular weight heparin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Patients will be evaluated for dose limiting toxicities until four weeks after combined radio-chemo-immunotherapy

SECONDARY OUTCOMES:
Metabolic response | After 6 weeks of chemo-immunotherapy
  Metabolic response, as measured by F-18-FDG PET-CT measurement of SUVmax
Secondary resectability | Decided by a multidisciplinary team 3-5 weeks after the end of neoadjuvant treatment
Major histopathological response rate | at surgery 4-6 weeks after end of neoadjuvant therapy
R-0 resection rate | at surgery 4-6 weeks after the end of neoadjuvant therapy
Surgical morbidity | within 30 days after surgery
Overall survival | Measured by median, 1-, 2-, and 3- year survival rates
Time to local and systemic progression after R0-resection | 5 years after completion of the trial treatement
Feasibility | Defined as completion of preoperative therapy (including surgery in patients with initially resectable tumors) and being alive 30 days postoperatively.
Toxicity (according to NCI-CTCAE, Version 4.0) | Within 30 days after completion of the trial treatement

CONTACTS AND LOCATIONS:
Overall Officials: Anna Dorothea Wagner, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland